CLINICAL TRIAL: NCT00961220
Title: A Phase I/II Multicenter Clinical Trial of O6Benzylguanine and Topical Carmustine in the Treatment of Refractory Early-Stage (IA-IIA) Cutaneous T-Cell Lymphoma
Brief Title: O6-Benzylguanine and Topical Carmustine in Treating Patients With Early-Stage IA-IIA Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02927; NCI-2012-02927 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 3405; CASE 3405-CC304 (Other: Case Comprehensive Cancer Center); 7080 (Other: CTEP); P30CA043703 (NIH); R21CA115057 (NIH); U01CA062502 (NIH)
Record Dates: First submitted 2009-08-16; First posted 2009-08-18 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Recurrent Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Stage I Mycosis Fungoides and Sezary Syndrome AJCC v7; Stage II Mycosis Fungoides and Sezary Syndrome AJCC v7
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Carmustine; carmustine, poliferprosan 20 drug combination; O(6)-benzylguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (O6-benzylguanine, carmustine) (Experimental): Patients receive O6-benzylguanine IV over 1 hour and apply topical carmustine to the total skin surface (excluding the lips, eyelids, and ulcerated lesions) 1 hour after completing O6-benzylguanine infusion on days 1-2. Treatment repeats every 2 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carmustine; Other: Laboratory Biomarker Analysis; Drug: O6-Benzylguanine

INTERVENTIONS:
Drug: Carmustine — Applied topically
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; Gliadel; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: O6-Benzylguanine — Given IV
  Other Names: 6-O-Benzylguanine; O(6)-Benzylguanine

SUMMARY:
This phase I/II trial studies the side effects and best dose of carmustine when given together with O6-benzylguanine and to see how well they work in treating patients with stage IA-IIA cutaneous T-cell lymphoma. Drugs used in chemotherapy, such as carmustine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. O6-benzylguanine may help carmustine work better by making cancer cells more sensitive to the drug. Giving O6-benzylguanine with carmustine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the cutaneous T-cell Lymphoma (CTCL) response rate and safety of O6BG (O6-benzylguanine) /BCNU (carmustine) when given biweekly as two consecutive daily doses.

SECONDARY OBJECTIVES:

I. To determine the laboratory correlates of clinical response and drug efficacy based upon O6-alkylguanine deoxyribonucleic acid (DNA) alkyltransferase (AGT) activity in CTCL lesions will be examined to determine the effects of consecutive day O6BG administration on the extent and duration of AGT depletion.

II. To determine the laboratory correlates of clinical response and drug efficacy based upon degree of induction of apoptosis and cell cycle arrest will be examined in the malignant T-cell population of lymphomatous tissue and in the constitutive cells of the skin to determine drug efficacy and toxicity through immunohistochemical techniques.

III. To determine the laboratory correlates of clinical response and drug efficacy based upon O-6-methylguanine-DNA methyltransferase (MGMT) gene mutations and changes in AGT expression will be examined as potential mechanisms for O6BG resistance in non-responding patients.

OUTLINE: This is a phase I, dose-escalation study of carmustine followed by a phase II study.

Patients receive O6-benzylguanine intravenously (IV) over 1 hour and apply topical carmustine to the total skin surface (excluding the lips, eyelids, and ulcerated lesions) 1 hour after completing O6-benzylguanine infusion on days 1-2. Treatment repeats every 2 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CTCL stages IA-IIA by histopathology and immunohistochemistry in screening biopsies confirmed at Case Western Reserve University within 6 months of enrollment; biopsies may be performed at the site of collaborating institutions and shipped to University Hospitals of Cleveland-Case Western Reserve University (UHC-CWRU)
* Performance status Eastern Cooperative Oncology Group (ECOG) grade 0, 1, or 2
* Patients must have recovered from toxicity of prior treatment and have received no CTCL therapy other than emollition for at least 4 weeks, with the exception of topical corticosteroids, which may be used up to 2 weeks before the trial start date
* Patients must have signed a consent form indicating the investigational nature of the treatment and its potential side effects
* White blood cell (WBC) at least 3.5 x10E9/L
* Absolute neutrophil count (ANC) at least 1.6 x10E9/L
* Platelets > 100,000/ul
* Bilirubin < 1.5 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT) within normal range
* Creatinine =< 1.5 mg/dL
* Electrolytes normal
* Controlled (diet and insulin) diabetes is permitted
* Demonstration of clinically normal lung function based on history and physical examination; patients with clinical evidence of pulmonary disease as determined by the investigator should have baseline lung function tests performed with demonstration of diffusing capacity of the lung for carbon monoxide (DLCO) >= 70%; a DLCO single breath, adjusted for hemoglobin, will be utilized; we will not use DLCO/alveolar volume (VA) for inclusion or exclusion in this study
* Patients must have cutaneous disease that is amenable to biopsy and must be willing to undergo several sequential biopsies
* Must have failed at least one conventional treatment for CTCL other than topical corticosteroids; this includes phototherapy, topical mechlorethamine, topical or oral bexarotene, radiation therapy, photopheresis, chemotherapy, and immunomodulatory agents such as interferon and other retinoids

Exclusion Criteria:

* Patients who have received prior treatment with topical or systemic BCNU or other nitrosoureas
* Patients with known central nervous system involvement or primary central nervous system (CNS) malignancies
* Patients with performance status ECOG grade 3 or 4
* Pregnant women, women who are breast feeding infants, or women with reproductive potential not practicing adequate contraception
* Patients with an active infection which requires hospitalization, or which may affect the patient?s safety if the patient was enrolled
* Patients with pulmonary disease as determined by history, physical examination, chest X-ray, or pulse oximetry with < 70% predicted DLCO
* CTCL patients with stage IIB-IVB disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2012-04-08 (Actual); Study Completion 2014-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Cooper, Principal Investigator — Case Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Henry Ford Hospital, Detroit, Michigan
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- [Derived] Tacastacas JD, Chan DV, Carlson S, Gerson SL, Dowlati A, Fu P, Lu K, Groft S, Rosenjack J, Honda K, McCormick TS, Cooper KD. Evaluation of O6-Benzylguanine-Potentiated Topical Carmustine for Mycosis Fungoides: A Phase 1-2 Clinical Trial. JAMA Dermatol. 2017 May 1;153(5):413-420. doi: 10.1001/jamadermatol.2016.5793. PMID 28199478

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from February 2010 to November 2013 from University Hospital Case Medical Center.
Groups:
- Treatment (O6-benzylguanine, Carmustine): Patients receive O6-benzylguanine IV over 1 hour and apply topical carmustine to the total skin surface (excluding the lips, eyelids, and ulcerated lesions) 1 hour after completing O6-benzylguanine infusion on days 1-2. Treatment repeats every 2 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  O6-benzylguanine: Given IV. 120 mg/m2 over 1 hour
  Carmustine (BCNU) will begin at a starting dose of 20 mg on Day 1. Beyond this first dose level, for each of the subsequent four patients enrolled, the BCNU dose will be escalated up to a limit of 40 mg total (given on day 1 only).
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Started | 17
Completed | 10
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 1
Not completed — No IV access for O6BG | 1
Not completed — O6BG no longer supplied | 1
Not completed — Complete Response prior to 12 courses | 1

BASELINE CHARACTERISTICS:
Population: Intention to treat
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Number analyzed (Participants) | 17
Age, Customized [Number; unit: participants]
  20-29 years | 2
  30-39 years | 5
  40-49 years | 4
  50-59 years | 2
  60-69 years | 3
  70-79 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Based on changes in modified SWAT assessment, patient responses will be classified as complete clinical response (CCR), partial response (PR), stable disease (SD), or progressive disease (PD). SWAT provides an accurate and reproducible assessment of cutaneous disease involvement based on body surface area of involvement and lesional thickness.
  CCR: No evidence of disease, 100% improvement for a duration of at least 4 weeks. PR: Greater than or equal to 50% decrease in SWAT score compared to baseline and improvement is maintained for at least 4 weeks. SD: Less than 50% decrease in SWAT score compared to baseline. PD: Increase of greater or equal to 25% of the SWAT score compared to baseline while the patient is actively taking the study drug
Time Frame: Up to 2 weeks after completion of study treatment
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Number analyzed (Participants) | 17
participants
  Complete Clinical Response-confirmed | 6
  Complete Clinical Response-unconfirmed | 2
  Partial Response | 8
  Progressive Disease | 1

2. Secondary Outcome: Changes in AGT (O6-alkylguanine DNA Alkyltransferase) Activity
Description: Examine AGT depletion at baseline, 24 hrs or 48 hrs, and 1 week after the first Infusion of O6BG. AGT levels will be determined by biochemical activity assay.
Time Frame: Baseline
Population: Attempts to stain AGT and caspase 3 were unsuccessful and there were no remaining tissues for other outcomes.
Groups:
- Treatment (O6-benzylguanine, Carmustine): Patients receive O6-benzylguanine IV over 1 hour and apply topical carmustine to the total skin surface (excluding the lips, eyelids, and ulcerated lesions) 1 hour after completing O6-benzylguanine infusion on days 1-2. Treatment repeats every 2 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  O6-benzylguanine: Given IV. 120 mg/m2 over 1 hour
  carmustine: Applied topically. BCNU will begin at a starting dose of 20 mg on Day 1. Beyond this first dose level, for each of the subsequent four patients enrolled, the BCNU dose will be escalated up to a limit of 40 mg total (given on day 1 only).
  laboratory biomarker analysis: Correlative studies
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Number analyzed (Participants) | 0

3. Secondary Outcome: Changes in AGT (O6-alkylguanine DNA Alkyltransferase) Activity
Description: as for outcome 2
Time Frame: 24 hours after the first infusion
Population: Attempts to stain AGT and caspase 3 were unsuccessful and there were no remaining tissues for other outcomes.
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Number analyzed (Participants) | 0

4. Secondary Outcome: Changes in AGT (O6-alkylguanine DNA Alkyltransferase) Activity
Description: as for outcome 2
Time Frame: 48 hours after the first infusion
Population: Attempts to stain AGT and caspase 3 were unsuccessful and there were no remaining tissues for other outcomes.
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Number analyzed (Participants) | 0

5. Secondary Outcome: Changes in AGT (O6-alkylguanine DNA Alkyltransferase) Activity
Description: as for outcome 2
Time Frame: 1 week after the first infusion
Population: Attempts to stain AGT and caspase 3 were unsuccessful and there were no remaining tissues for other outcomes.
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Number analyzed (Participants) | 0

6. Secondary Outcome: Changes in the Apoptosis
Description: Comparing skin biopsy specimens of BCNU-protected CTCL lesional specimens vs BCNU-treated lesional specimens at 24 hours, using immunohistochemical staining for Ki-67, PCNA, bcl-2, and caspase-3, as well as y2HAX and TUNEL assays. The apoptotic index will be calculated from these results.
Time Frame: at 24 hours after the first infusion
Population: Attempts to stain AGT and caspase 3 were unsuccessful and there were no remaining tissues for other outcomes.
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Number analyzed (Participants) | 0

7. Secondary Outcome: Changes in the Apoptosis
Description: Comparing skin biopsy specimens of BCNU-protected CTCL lesional specimens vs BCNU-treated lesional specimens at 48 hours, using immunohistochemical staining for Ki-67, PCNA, bcl-2, and caspase-3, as well as y2HAX and TUNEL assays. The apoptotic index will be calculated from these results.
Time Frame: at 48 hours after the first infusion
Population: Attempts to stain AGT and caspase 3 were unsuccessful and there were no remaining tissues for other outcomes.
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Number analyzed (Participants) | 0

8. Secondary Outcome: Changes in the Cell Cycle/Proliferation
Description: Comparing skin biopsy specimens of BCNU-protected CTCL lesional specimens vs BCNU-treated lesional specimens at 24 hours, using immunohistochemical staining for Ki-67, PCNA, bcl-2, and caspase-3, as well as y2HAX and TUNEL assays. The proliferation rate will be calculated from these results.
Time Frame: at 24 hours after the first infusion
Population: Attempts to stain AGT and caspase 3 were unsuccessful and there were no remaining tissues for other outcomes.
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Number analyzed (Participants) | 0

9. Secondary Outcome: Changes in the Cell Cycle/Proliferation
Description: Comparing skin biopsy specimens of BCNU-protected CTCL lesional specimens vs BCNU-treated lesional specimens at 48 hours, using immunohistochemical staining for Ki-67, PCNA, bcl-2, and caspase-3, as well as y2HAX and TUNEL assays. The proliferation rate will be calculated from these results.
Time Frame: at 48 hours after the first infusion
Population: Attempts to stain AGT and caspase 3 were unsuccessful and there were no remaining tissues for other outcomes.
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Number analyzed (Participants) | 0

10. Secondary Outcome: Changes in DNA Damage- Cytotoxicity
Description: Immunohistochemistry will be used to assess expression of these proteins in keratinocytes, epidermal lymphocytes, and dermal lymphocytes, to determine the effects of BCNU cytotoxicity in each subpopulation of cells
Time Frame: 24 hours after the first infusion
Population: Attempts to stain AGT and caspase 3 were unsuccessful and there were no remaining tissues for other outcomes.
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Number analyzed (Participants) | 0

11. Secondary Outcome: Changes in DNA Damage- Cytotoxicity
Description: as for outcome 10
Time Frame: 48 hours after the first infusion
Population: Attempts to stain AGT and caspase 3 were unsuccessful and there were no remaining tissues for other outcomes.
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Number analyzed (Participants) | 0

12. Secondary Outcome: Changes in AGT Inactivation in Non-responding Patients
Description: Changes in AGT levels will be determined by biochemical activity assay from first course to seventh course of treatment.
Time Frame: After first course at 2 weeks
Population: Attempts to stain AGT and caspase 3 were unsuccessful and there were no remaining tissues for other outcomes.
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Number analyzed (Participants) | 0

13. Secondary Outcome: Changes in AGT Inactivation in Non-responding Patients
Description: Changes in AGT levels will be determined by biochemical activity assay from first course to seventh course of treatment.
Time Frame: After seventh course at 14 weeks
Population: Attempts to stain AGT and caspase 3 were unsuccessful and there were no remaining tissues for other outcomes.
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from during treatment over a 6 month time period.
Arm/Group | Treatment (O6-benzylguanine, Carmustine)
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 16/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (O6-benzylguanine, Carmustine) (N=17)
ACNEIFORM RASH (Skin and subcutaneous tissue disorders) | 1
ALKALINE PHOSPHATASE ELEVATED (Investigations) | 1
ANEMIA (Blood and lymphatic system disorders) | 3
BLOATING (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
CREATININE ELEVATION (Investigations) | 1
CUTANEOUS HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 12
DIZZINESS (Nervous system disorders) | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 2
FATIGUE (General disorders) | 10
GLUCOSE LOW (Metabolism and nutrition disorders) | 1
HEADACHE (Nervous system disorders) | 8
INJECTION SITE REACTION or PAIN (General disorders) | 2
JOINT PAINS (Musculoskeletal and connective tissue disorders) | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 1
MONOCYTE ELEVATION (Blood and lymphatic system disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1
NAUSEA (Gastrointestinal disorders) | 8
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 9
PRURITUS (Skin and subcutaneous tissue disorders) | 9
RASH/ DESQUAMATION (Skin and subcutaneous tissue disorders) | 11
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 1
TELANGIECTASIA (Skin and subcutaneous tissue disorders) | 1
TOTAL BILIRUBIN ELEVATED (Investigations) | 1
TRANSAMINASE ELEVATION (Investigations) | 9
URIC ACID ELEVATION (Renal and urinary disorders) | 2
URINE SPECIFIC GRAVITY ELEVATED (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less